CLINICAL TRIAL: NCT07315516
Title: The Effects of Natural Bioactive Compounds on Sleep and Stress: A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Sleep and Stress Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Gencor Pacific Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVESLE
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Sleep Disorder (Disorder); Stress; Anxiety
Keywords: Sleep complaints
MeSH Terms: conditions — Sleep Wake Disorders; Anxiety Disorders | interventions — lavender oil; palmidrol; oleoylethanolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CPO Lavender oil (Experimental): 85mg CPO Lavender oil will be administered daily, This will be taken as a capsule, 1 capsule daily for 57 days.
  Interventions: Dietary Supplement: Lavender Oil
- Levagen+ PEA (Experimental): 75mg Levagen+ PEA will be administered daily, This will be taken as a capsule, 1 capsule daily for 57 days.
  Interventions: Dietary Supplement: Palmitoylethanolamide (PEA)
- Trpti OEA (Experimental): 150mg Trpti OEA will be administered daily, This will be taken as a capsule, 1 capsule daily for 57 days.
  Interventions: Dietary Supplement: Oleoylethanolamide
- Placebo (Placebo Comparator): A placebo capsule containing microcrystalline cellulose will be taken daily, 1 capsule will be taken each day for 57 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lavender Oil — 85mg CPO Lavender oil will be administered daily. This will be taken as a capsule, 1 capsule daily for 57 days.
  Other Names: CPO Lavender oil
  Arms: CPO Lavender oil
Dietary Supplement: Palmitoylethanolamide (PEA) — 75mg Levagen+ PEA will be administered daily. This will be taken as a capsule, 1 capsule daily for 57 days.
  Other Names: Levagen+
  Arms: Levagen+ PEA
Dietary Supplement: Oleoylethanolamide — 150mg Trpti OEA will be administered daily. This will be taken as a capsule, 1 capsule daily for 57 days
  Other Names: Trpti
  Arms: Trpti OEA
Other: Placebo — A placebo capsule containing microcrystalline cellulose will be taken daily, 1 capsule will be taken each day for 57 days.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if natural supplements (lavender oil, PEA, and OEA) work to improve sleep and reduce stress in adults with moderate stress levels and sleep difficulties. It will also learn about the safety of these natural supplements.

The main questions it aims to answer are:

* Do these supplements improve sleep quality?
* Do they reduce perceived stress levels?
* Do they reduce anxiety symptoms?
* What medical problems do participants have when taking these supplements?

Researchers will compare three active treatment groups (lavender oil, PEA, Trpti which contains OEA) to a placebo (a look-alike capsule that contains no active ingredients) to see if these natural supplements work to improve sleep and reduce stress.

Participants will take 1 capsule (either active supplement or placebo) every day for 8 weeks and attend 2 clinic visits with a phone check in in between.

DETAILED DESCRIPTION:
The Effects of Natural Bioactive Compounds on Sleep and Stress: A Randomized Double-Blind Placebo-Controlled Trial This four-arm, parallel-group trial evaluates bioactive compounds targeting stress-sleep pathophysiology (lavender oil, PEA, and OEA). The 8-week intervention employs validated psychometric instruments alongside salivary biomarkers providing objective HPA axis and circadian rhythm assessment. The trial enrolls 240 participants (60 per arm) with moderate stress (PSS ≥14) and sleep complaints.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adults aged 18 and over.
* Able to provide informed consent.
* Score of at least 14 on the Perceived Stress Scale (PSS).
* Those with a sleep complaint with a frequency of at least 2 times per week(1)
* Agree not to use other dietary supplements for sleep, depression, stress or anxiety other than the investigational product during entire study period.
* Agree not to change current diet and/or exercise frequency or intensity during entire study period.
* Agree to not participate in another clinical trial during the study period.

  1. Sleep complaints are defined as difficulty initiating sleep, or difficulty maintaining sleep, or early-morning awakening with inability to return to sleep and causing distress or impairment in social, occupational, educational, academic, behavioural, or other important areas of functioning.)

Exclusion Criteria:

* A WHO-5 Well-Being Index score ≤ 28
* Those with severe sleep complaints (Insomnia Severity Index >21)
* Taking prescribed sleep, depression or anxiety medication
* Have a serious illness e.g. asthma, depression, anxiety disorder, bipolar disorder, insomnia, organic sleep disorders (i.e. sleep apnoea), neurological disorders such as MS, kidney disease, liver disease or heart conditions
* Have an unstable illness e.g. diabetes and thyroid gland dysfunction
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy including low dose aspirin
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>21 alcoholic drinks week)
* Those consuming more than 500mg caffeine per day
* Pregnant or lactating women
* Allergic to any of the ingredients in active or placebo formula
* Participants who are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 1 month
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Perceived stress via Perceived Stress Scale (PSS) | Day 1 to day 57
  Change from baseline to the end of the study period in Perceived stress via Perceived Stress Scale (PSS). The Perceived Stress Scale is a self-reported tool for measuring psychological stress. A total PSS-10 score from 0 to 40 is presented, with higher scores representing higher levels of stress.
Anxiety via Beck Anxiety Inventory (BAI) | Day 1 to day 57
  Change from baseline to the end of the study period in Anxiety via Beck Anxiety Inventory (BAI). The BAI is a 21-item self-report questionnaire evaluating anxiety symptoms, rated on a 4-point scale.
Sleep quality | Day 1 to day 57
  Change from baseline to the end of the study period in Sleep quality. This will be measured via Pittsburgh Sleep Quality Index (PSQI) and Consensus Sleep Diary. The PSQI is a self-report questionnaire used to evaluate overall sleep quality. Each of the 19 items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The Consensus Sleep Diary is designed to gather information about daily sleep patterns.

SECONDARY OUTCOMES:
Mental wellbeing | Day 1 to day 57
  Change from baseline to the end of the study period in Mental wellbeing via The World Health Organization-Five Well-Being Index (WHO-5). The WHO-5 is a self-report instrument measuring mental well-being. It consists of five statements relating to the past two weeks. Each statement is rated on a 6-point scale, with higher scores indicating better mental well-being. A score ≤ 50 (or < 13 in the raw score) is associated with poor well-being or psychological distress and a score ≤ 28 may denote possible clinical symptoms of depression.
Mood | Day 1 to day 57
  Change from baseline to the end of the study period in Mood via Profile of mood states (POMS). The POMS is a self-reported questionnaire consisting of 65 items, designed to evaluate individuals within seven different mood domains: fatigue-inertia, anger-hostility, vigor-activity, confusion-bewilderment, depression-dejection, tension-anxiety, and friendliness.
Sleep duration | Day 1 to day 57
  Change from baseline to the end of the study period in Sleep duration via PSQI and Consensus Sleep Diary. The PSQI is a self-report questionnaire used to evaluate overall sleep quality. Each of the 19 items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The Consensus Sleep Diary is designed to gather information about daily sleep patterns.
Sleep onset latency | Day 1 to day 57
  Change from baseline to the end of the study period in Sleep onset latency as measured by duration of time (minutes) from turning light off to falling asleep (PSQI and Consensus Sleep Diary). The PSQI is a self-report questionnaire used to evaluate overall sleep quality. Each of the 19 items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The Consensus Sleep Diary is designed to gather information about daily sleep patterns.
Sleep efficiency | Day 1 to day 57
  Change from baseline to the end of the study period in Sleep efficiency as measured by ratio of total sleep time to time in bed (PSQI). The PSQI is a self-report questionnaire used to evaluate overall sleep quality. Each of the 19 items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Daytime sleepiness | Day 1 to day 57
  Change from baseline to the end of the study period in Daytime sleepiness via Functional Outcomes of Sleep Questionnaire (FOSQ-10). The FOSQ-10 consists of 10 items distributed among 5 subscales i.e. general productivity (2 item), activity level (3 items), vigilance (3 items), social outcomes (1 item) and sexual relationship (1 item). Items are rated on a scale of 1-4 (1 = extreme difficulty, 2 = moderate difficulty, 3 = a little difficulty, 4 = no difficulty). The total score is the sum of the 5 sub scores.
Eating in response to experienced stress | Day 1 to day 57
  Change from baseline to the end of the study period in Eating in response to experienced stress via the Salzburg Stress Eating Scale (SSES). The SSES is a questionnaire use to measure eating in response to experienced stress. The response categories range from 'I eat much less than usual' to 'I eat much more than usual' and are scored on a 5-point Likert scale, i.e., a score from 1 - 5. Higher scores indicate that the respondent eats more when stressed is experienced.
Serotonin | Day 1 to day 57
  Change from baseline to the end of the study period in serotonin via saliva test.
Cortisol | Day 1 to day 57
  Change from baseline to the end of the study period in cortisol via saliva test.
Melatonin | Day 1 to day 57
  Change from baseline to the end of the study period in melatonin via saliva test.
Safety via AE monitoring | Day 1 to day 57
  Change from baseline to the end of the study period in Safety via AE monitoring
Safety via vital signs (blood pressure) | Day 1 to day 57
  Change from baseline to the end of the study period in safety via vital signs (blood pressure).
Safety via vital signs (heart rate) | Day 1 to day 57
  Change from baseline to the end of the study period in safety via vital signs (heart rate).
Safety via vital signs (O2 saturation) | Day 1 to day 57
  Change from baseline to the end of the study period in safety via vital signs (O2 saturation).
Safety via vital signs (temperature) | Day 1 to day 57
  Change from baseline to the end of the study period in safety via vital signs (temperature).

CONTACTS AND LOCATIONS:
Overall Officials: RV Venkatesh, Study Director — Gencor Pacific
Locations (1):
- RDC Clinical, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: Undecided